CLINICAL TRIAL: NCT04212000
Title: A Phase 1 Randomized, Open-Label, Two-Period,Two-Sequence Crossover Study to Evaluate the Relative Oral Bioavailability of Levoketoconazole and Ketoconazole Tablets in Healthy Subjects
Brief Title: Bioavailability of Levoketoconazole and Ketoconazole Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cortendo AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LKC101A
Record Dates: First submitted 2019-12-11; First posted 2019-12-26 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levoketoconazole (Experimental): Levoketoconazole 150 mg
  Interventions: Drug: Levoketoconazole
- Ketoconazole (Active Comparator): Ketoconazole 200 mg
  Interventions: Drug: Ketoconazole

INTERVENTIONS:
Drug: Levoketoconazole — Levoketoconazole tablet
  Other Names: COR-003
  Arms: Levoketoconazole
Drug: Ketoconazole — Ketoconazole tablet
  Arms: Ketoconazole

SUMMARY:
This is a phase 1, randomized, open-label, single-dose, two-period, two-sequence crossover study in healthy male and female subjects to evaluate the relative oral bioavailability of levoketoconazole tablets (the test drug) and ketoconazole tablets (the reference drug product).

DETAILED DESCRIPTION:
This is a phase 1, randomized, open-label, single-dose, two-period, two-sequence crossover study in healthy male and female subjects to evaluate the relative oral bioavailability of levoketoconazole tablets (the test drug) and ketoconazole tablets (the reference drug product). Subjects will be randomized to receive a single oral dose of 150 mg levoketoconazole (Study Drug A) or a single oral dose of 200 mg ketoconazole (Study Drug B) in each period.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 55 years of age, inclusive, at time of consent.
2. Body mass index (BMI) between 18.0 and 32.0 kg/m2,inclusive.
3. In good general physical health as determined by absence of clinically significant medical history, physical examination findings, vital signs, clinical laboratory evaluations, and ECG measurements.
4. Has not consumed and agrees to abstain from taking any prescription drugs, dietary supplements including vitamins and herbal preparations, or non-prescription drugs for 14 days prior to clinical research unit (CRU) admission, during washout period, and through Follow-Up.
5. Has not consumed alcohol-containing beverages for 3 days prior to CRU admission and agrees not to consume alcohol through Follow-Up.
6. Is a nonsmoker (for at least 3 months) with negative urinary cotinine test at Screening and agrees to abstain from tobacco-and nicotine-containing products for the duration of the study.

Exclusion Criteria:

1. Evidence of any out-of-normal-range laboratory value at Screening that has not been reviewed, approved, and documented as Not Clinically Significant by the Investigator.
2. Concurrent medical illness that would interfere with the conduct of the study in the opinion of the Investigator.
3. History or presence of clinically significant cardiovascular, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, psychiatric, renal, hepatic, chronic respiratory, or gastrointestinal disease as judged by the Investigator.
4. Positive urine drug screen for drugs-of-abuse, including cocaine, tetrahydrocannabinol, opioids, benzodiazepines, amphetamines, and barbiturates,and/or positive urine screen for alcohol at Screening and CRU admission.
5. Treatment with an investigational drug within the longer of 30 days or five half-lives of the investigational drug preceding the first dose of study drug.
6. Positive for HIV, hepatitis B, and/or hepatitis C on Screening assessments.
7. Acute illness within 7 days of CRU admission.
8. Donated plasma within 7 days of drug administration.
9. Donated 1 or more pints of blood (or equivalent blood loss) within 30 days prior to drug administration.
10. History of caffeine consumption exceeding 8 cups coffee/day within 14 days prior to first dose, or consumption of any caffeine-or chocolate-containing products for 3 days prior to CRU admission each week.
11. Female subjects who are pregnant or lactating.
12. Males with hemoglobin less than 12.0 g/dL at Screening or CRU admission; Females with hemoglobin less than 11.0 g/dL at Screening or CRU admission
13. Had difficulties with swallowing whole tablets.
14. Body habitus preventing repeated venipuncture as required by protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Ratio of geometric least squares means for AUClast of plasma levoketoconazole (2S,4R-ketoconazole) | 24 hours
  Point estimates and 90 percent (%) confidence intervals (CIs) for the dose-normalized ratios of geometric least squares means between Test (levoketoconazole) and Reference (ketoconazole)
Ratio of geometric least squares means for AUCinf of plasma levoketoconazole (2S,4R-ketoconazole) | 24 hours
  Point estimates and 90 percent (%) confidence intervals (CIs) for the dose-normalized ratios of geometric least squares means between Test (levoketoconazole) and Reference (ketoconazole)
Ratio of geometric least squares means for Cmax of plasma levoketoconazole (2S,4R-ketoconazole) | 24 hours
  Point estimates and 90 percent (%) confidence intervals (CIs) for the dose-normalized ratios of geometric least squares means between Test (levoketoconazole) and Reference (ketoconazole)

SECONDARY OUTCOMES:
Terminal phase rate constant (λz) | 24 hours
  Single-dose plasma PK parameters after a single administration of levoketoconazole and ketoconazole in the fasted state including λz
Time to Maximum Plasma concentration (Tmax) | 24 hours
  Single-dose plasma PK parameters after a single administration of levoketoconazole and ketoconazole in the fasted state including Tmax
Lag-time (Tlag) | 24 hours
  Single-dose plasma PK parameters after a single administration of levoketoconazole and ketoconazole in the fasted state including: Tlag
Apparent systemic clearance (CL/F) | 24 hours
  Single-dose plasma PK parameters after a single administration of levoketoconazole and ketoconazole in the fasted state including: CL/F
The percentage of area under the plasma concentration-time curve extrapolated from time 0 to infinity as a percentage of total AUC (%AUCext) | 24 hours
  Single-dose plasma PK parameters after a single administration of levoketoconazole and ketoconazole in the fasted state including: %AUCext
Volume of Distribution (Vz/F) | 24 hours
  Single-dose plasma PK parameters after a single administration of levoketoconazole and ketoconazole in the fasted state including: Vz/F
Elimination half-life (T1/2) | 24 hours
  Single-dose plasma PK parameters after a single administration of levoketoconazole and ketoconazole in the fasted state including: t½
Incidence of adverse events (AEs) | 35 days
  Incidence of Treatment-Emergent AEs (TEAEs), AEs of special interest, and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Valencia, MD, Study Director — Cortendo AB
Locations (1):
- Pharmaceutical Research Associates, Inc., Salt Lake City, Utah, United States